CLINICAL TRIAL: NCT02516774
Title: A Phase I Trial Assessing Adalimumab (Humira®), a Tumor Necrosis Factor α Inhibitor Combined to Chemotherapy and Radiotherapy in Patients With Anaplastic Thyroid Cancers
Brief Title: A Trial of Adalimumab Combined to Chemotherapy and Radiotherapy in Patients With Anaplastic Thyroid Cancers
Acronym: TAM-RT
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No patients enrolled
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-002618-22; 2014/2142 (Other: CSET number)
Record Dates: First submitted 2015-04-29; First posted 2015-08-06 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Anaplastic Thyroid Cancers
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose escalation (Experimental): Adalimumab will be administrated subcutaneously 1h prior to chemotherapy at D1W1, D1W3, D1W5, D1W7, and D1W9, starting with the chemotherapy for a total duration of 9 weeks (5 injections in total)
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab
  Other Names: Humira®

SUMMARY:
The hypothesis is that the particular richness of ATC's microenvironment in TAMs creates a unique opportunity for using Tumor Necrosis Factor blockade during chemotherapy and radiotherapy in order to counteract tumor resistance to therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven anaplastic thyroid cancers (localized or metastatic)
2. Life-expectancy > 12 weeks
3. No previous treatment for anaplastic thyroid cancer excepted surgery or crizotinib
4. Written Informed consent signed
5. Age > 18 years
6. WHO 0-3
7. Neutrophil count > 1500 /mm3, Haemoglobin > 9 gr/dL, Platelet count > 100,000/mm3
8. Bilirubin < 1.5 mg/dL, Transaminases < 3 N in absence of liver metastases or <5 N if presence of liver metastases, PT > 70%
9. Creatinine clearance > 50ml/mn (calculated by the MDRD formula)
10. Negative pregnancy test in women of childbearing potential within 14 days prior to treatment initiation (premenopausal or less than 12 months of amenorrhea post-menopause, and who have not undergone surgical sterilization). Both men and women (of childbearing potential) who are sexually active, must use adequate contraception, during and for at least 6 months post-treatment.
11. Evaluable disease > 1 cm within the cervico-mediastinal field of radiotherapy according to the Response Evaluation Criteria in Solid Tumors 1.1 criteria
12. Patient affiliated to social security regimen or beneficiary of such regimen

Exclusion Criteria:

1. Prior treatment with anthracyclines
2. Left Ventricular Ejection Fraction (LVEF) < 50%
3. Known allergy to Adalimumab, doxorubicin, cisplatin, carboplatin or paclitaxel
4. Chronic or acute infection < 15 days
5. Pregnant or breastfeeding patients
6. Any other malignancy in the past 5 years except basal cell carcinoma and carcinoma in situ of the cervix
7. Previous and/or active demyelinating disease, such as multiple sclerosis
8. Prior radiotherapy to the neck
9. Concomitant therapy with agents otherwise used in the treatment of cancer (for example methotrexate for rheumatoid arthritis)
10. Chronic (> 3 months) treatment with oral corticosteroids or another immunosuppressant within 15 days prior registration
11. Patients with an active bleeding diathesis or taking an oral vitamin K antagonist (except low-dose Coumadin (warfarin sodium))
12. Other concurrent severe and/or uncontrolled disease which could compromise participation in the study (i.e. uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, unstable angina, or congestive heart failure - New York Heart Association Class III or IV, ventricular arrhythmia, active ischemic heart disease, myocardial infarction during the previous six months, chronic liver or renal disease, active upper GI tract ulceration)
13. Patient already enrolled in another therapeutic trial involving an investigational substance, and when such a substance has been taken during the previous 4 weeks
14. Chronic Hepatitis B virus and previous viral hepatitis with risk of reactivation, Hepatitis C virus and human immunodeficiency virus 1 or human immunodeficiency virus 2 infection, active or latent tuberculosis infection
15. Persons deprived of their freedom or under guardianship, or for whom it would be impossible to undergo the medical follow-up required by the trial, for geographic, social or psychological reasons Refusal or absence of biopsy (excepted for initial pathological diagnosis) will not constitute an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Recommended dose | Up to 9 weeks
  Two dose levels will be investigated :
  * Level 1: 20 mg at D1W1, D1W3, D1W5, D1W7 and D1W9.
  * Level 2: 40 mg at D1W1, D1W3, D1W5, D1W7 and D1W9.

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val de Marne, France